CLINICAL TRIAL: NCT03037307
Title: A Bite Force Study Assessing Two Currently Marketed Denture Adhesive Products Compared to No-Adhesive Control
Brief Title: A Clinical Bite Force Study of Two Marketed Adhesives Against no Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 207545
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-04

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (Experimental): Participants will topically apply the test product to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
  Interventions: Other: Test Product
- Positive Control (Active Comparator): Participants will topically apply the positive control to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
  Interventions: Other: Positive Contol
- Negative Control (Other): Participants of this group will not be assigned to any treatment.
  Interventions: Other: Negative Control

INTERVENTIONS:
Other: Test Product — Five strips of test adhesive cream for upper denture, as per application instructions.
  Arms: Test product
Other: Positive Contol — Three dabs of positive control adhesive cream for upper denture, as per application instructions.
  Arms: Positive Control
Other: Negative Control — No adhesive
  Arms: Negative Control

SUMMARY:
The objective of this study will be to compare bite force (BF) measurements over a 12-hour period of a currently marketed denture adhesive cream based on carbomer technology (test), with a positive control and a negative/no treatment control.

DETAILED DESCRIPTION:
This will be a single centre, randomized, crossover, 3-treatment, 3-period study to compare BF measurements over a 12 hour period of a currently marketed denture adhesive cream based on carbomer technology (test), with a positive control, and a negative/no treatment control. A short questionnaire regarding the flavor and texture characteristics of each denture adhesive after a single use will also be used to generate data for these attributes. This study included four visits: Visit 1 (screening visit), Visit 2, 3, 4 (treatment visits).

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 to 85 years.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination; absence of any condition that could affect the participant's safety or wellbeing or their ability to understand and follow study procedures and requirements.
* Diagnosis: a) Completely edentulous maxillary arch restored with a conventional full acrylic based upper complete denture, b) Dentate, partial or full edentulous mandibular arch. Partial or full edentulous arch may be restored with a stable complete, partial or implant supported denture, c) Maxillary dentures must be considered to be moderately well-fitting at the screening visit (Kapur Index, Olshan Modification: retention score >2, stability score >2) d) Maxillary dentures and mandibular dentures, if present, must be considered to be well-made based on design and construction criteria specified in the protocol e) The qualifying maxillary incisal BF readings (without adhesive) must be less than or equal to 9 pounds at the Screening Visit and subsequent visit pretreatment baseline bites. f) At least 2 of the 4 qualifying bite readings at the Screening Visit must be reproducible (+2lb). At subsequent visits the bite force readings must be within +2lb for 1 of the 3 practice bites and the pre-treatment baseline bite.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* A woman who is known to be pregnant or who is intending to become pregnant (self-reported) over the duration of the study.
* A woman who is breast-feeding.
* a) Implanted with a cardiac pacemaker, b) Daily doses of medication that might interfere with the ability to perform the study according to protocol (as determined by the Investigator), c) Insulin dependent diabetics, d) Taking or have taken a bisphosphonate drug for treatment of osteoporosis, e) A serious chronic disease requiring hospitalization, f) Any condition not previously mentioned that in the Investigator's opinion may impair the study evaluation.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* a) Any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the participant's participation in the study, b) Any participant clinically identified as having an incisal bite relation which could affect the bite force measurements, c) Severe dry mouth that may affect denture retention in the opinion of the Investigator, d) OST examination findings such as stomatitis, open sores, lesions, redness or swelling that, in the opinion of the investigator, could affect the participant's participation in the study. e) A serious chronic disease requiring hospitalization. f) Any condition not previously mentioned that in the Investigator's opinion may impair the study evaluation.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* a) Any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the participant's participation in the study, b) Any participant clinically identified as having an incisal bite relation which could affect the bite force measurements, c) Severe dry mouth that may affect denture retention in the opinion of the Investigator, d) OST examination findings such as stomatitis, open sores, lesions, redness or swelling that, in the opinion of the investigator, could affect the participant's participation in the study.
* a) Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit, b) Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* A participant who is unwilling to refrain from smoking, including e-cigarettes and the use of chewing tobacco or other tobacco products for the duration of screening and each treatment day (12-14 hours).
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Varghese R, Burnett GR, Souverain A, Patil A, Gossweiler AG. A randomised bite force study assessing two currently marketed denture adhesive products compared with no-adhesive control. Clin Exp Dent Res. 2019 May 14;5(3):276-283. doi: 10.1002/cre2.182. eCollection 2019 Jun. PMID 31249709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in the United States.
Pre-assignment Details: A total of 53 participants were screened. Out of which 44 participants were randomized in the study. 9 participants were not randomized because they did not meet the study criteria.
Groups:
- Test Adhesive/No Treatment/Positive Control Adhesive: Participants in this arm received topical application of test adhesive, followed by no treatment, positive control adhesive in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products were applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- Test Adhesive/Positive Control Adhesive/No Treatment: Participants in this arm received topical application of test adhesive, followed by positive control adhesive and no treatment in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products was applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- No Treatment/Test Adhesive/Positive Control Adhesive: Participants in this arm received no treatment, followed by topical application of test adhesive and positive control adhesive in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products was applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- No Treatment/Positive Control Adhesive/Test Adhesive: Participants in this arm received no treatment, followed by topical application of positive control adhesive and test adhesive in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products was applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- Positive Control Adhesive/Test Adhesive/No Treatment: Participants in this arm received topical application of positive control adhesive, followed by test adhesive and no treatment in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products was applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- Positive Control Adhesive/No Treatment/Test Adhesive: Participants in this arm received topical application of positive control adhesive, followed by no treatment and test adhesive in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of at least 24 hours up to 14 days. Study products was applied by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
Period: Period 1
Arm/Group | Test Adhesive/No Treatment/Positive Control Adhesive | Test Adhesive/Positive Control Adhesive/No Treatment | No Treatment/Test Adhesive/Positive Control Adhesive | No Treatment/Positive Control Adhesive/Test Adhesive | Positive Control Adhesive/Test Adhesive/No Treatment | Positive Control Adhesive/No Treatment/Test Adhesive
Started | 7 | 7 | 8 | 7 | 7 | 8
Completed | 7 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did Not Meet Study Criteria | 0 | 0 | 0 | 1 | 0 | 0
Period: Wash Out Period 1
Arm/Group | Test Adhesive/No Treatment/Positive Control Adhesive | Test Adhesive/Positive Control Adhesive/No Treatment | No Treatment/Test Adhesive/Positive Control Adhesive | No Treatment/Positive Control Adhesive/Test Adhesive | Positive Control Adhesive/Test Adhesive/No Treatment | Positive Control Adhesive/No Treatment/Test Adhesive
Started | 7 | 7 | 8 | 6 | 7 | 8
Completed | 7 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Test Adhesive/No Treatment/Positive Control Adhesive | Test Adhesive/Positive Control Adhesive/No Treatment | No Treatment/Test Adhesive/Positive Control Adhesive | No Treatment/Positive Control Adhesive/Test Adhesive | Positive Control Adhesive/Test Adhesive/No Treatment | Positive Control Adhesive/No Treatment/Test Adhesive
Started | 7 | 7 | 8 | 6 | 7 | 8
Completed | 7 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out Period 2
Arm/Group | Test Adhesive/No Treatment/Positive Control Adhesive | Test Adhesive/Positive Control Adhesive/No Treatment | No Treatment/Test Adhesive/Positive Control Adhesive | No Treatment/Positive Control Adhesive/Test Adhesive | Positive Control Adhesive/Test Adhesive/No Treatment | Positive Control Adhesive/No Treatment/Test Adhesive
Started | 7 | 7 | 8 | 6 | 7 | 8
Completed | 7 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test Adhesive/No Treatment/Positive Control Adhesive | Test Adhesive/Positive Control Adhesive/No Treatment | No Treatment/Test Adhesive/Positive Control Adhesive | No Treatment/Positive Control Adhesive/Test Adhesive | Positive Control Adhesive/Test Adhesive/No Treatment | Positive Control Adhesive/No Treatment/Test Adhesive
Started | 7 | 7 | 8 | 6 | 7 | 8
Completed | 7 | 7 | 8 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: All randomized participants who received test adhesive, positive control adhesive and did not receive any treatment were included in the baseline assessment.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for the Incisal Bite Force (Positive Control Adhesive Versus [vs.] Negative Control)
Description: Area over baseline over 12 hours (AOB0-12) was assessed to measure the incisal bite force. AOB0-12 was calculated as area under the curve over 12 hours [AUC0-12])/12 hours minus baseline bite force (pounds [lbs]). AUC0-12 was calculated using the trapezoidal method. This transformation returned the measurement to the same scale as the original observations. Higher values of AOB0-12 demonstrate a stronger bite force overtime than lower values.
Time Frame: Up to 12 hours
Population: Analysis for this outcome was performed on intention-to-treat (ITT) population which included all randomized participants with at least one post baseline assessment of efficacy.
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Positive Control Adhesive: Participants of this arm received topical application of positive control adhesive (super poligrip free, commercially available) by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
- Negative Control: Participants of this arm did not receive any adhesive to apply on upper denture.
Arm/Group | Positive Control Adhesive | Negative Control
Number analyzed (Participants) | 44 | 44
lbs | 4.78 (0.657) | 2.03 (0.657)
Statistical Analysis 1: Comparison: Positive Control Adhesive vs Negative Control; Test type: Other; p < .0001, ANCOVA — Treatment Comparison for study validity; ANCOVA: factors for participant (random effect); period & treatment, participant-level & period-level pre-treatment baseline bite force as covariates; Least square (LS) mean difference = 2.76, 95% CI 2-sided [1.89 to 3.63] — Difference is first-named treatment minus second-named treatment such that a positive difference favours the first named treatment

2. Primary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for the Incisal Bite Force (Test Adhesive vs. Negative Control)
Description: Area over baseline over 12 hours (AOB0-12) was assessed to measure the incisal bite force. AOB0-12 was calculated as area under the curve over 12 hours [AUC0-12])/12 hours minus baseline bite force (lbs). AUC0-12 was calculated using the trapezoidal method. This transformation returned the measurement to the same scale as the original observations. Higher values of AOB0-12 demonstrate a stronger bite force overtime than lower values.
Time Frame: Up to 12 hours
Population: Analysis for this outcome was performed on ITT population which included all randomized participants with at least one post baseline assessment of efficacy.
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Test Adhesive: Participants of this arm received topical application of test adhesive (commercially available) by site study staff, to clean wet denture (upper denture) fit surface in a pattern consistent with product label and application instructions.
Arm/Group | Test Adhesive | Negative Control
Number analyzed (Participants) | 44 | 44
lbs | 4.15 (0.659) | 2.03 (0.657)
Statistical Analysis 1: Comparison: Test Adhesive vs Negative Control; Test type: Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) mean difference = 2.12, 95% CI 2-sided [1.25 to 3.00] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 51 days (AEs were collected from OST examination from screening until 5 days following last administration of study product on Visit 4)
Groups:
- Overall Participants: This arm included all the participants randomized to receive test adhesive, positive control adhesive and no treatment.
Arm/Group | Test Adhesive | Positive Control Adhesive | Negative Control | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 2/42 | 2/43 | 0/44 | 4/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Adhesive (N=42) | Positive Control Adhesive (N=43) | Negative Control (N=44) | Overall Participants (N=44)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03037307/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT03037307/SAP_001.pdf